CLINICAL TRIAL: NCT00000627
Title: Pilot Study to Determine the Feasibility of Fluconazole for Induction Treatment and Suppression of Relapse of Histoplasmosis in Patients With the Acquired Immunodeficiency Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 174; R-0245; 11149 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Histoplasmosis
Keywords: Pilot Projects; Histoplasmosis; Drug Evaluation; Fluconazole; Acquired Immunodeficiency Syndrome; Recurrence
MeSH Terms: conditions — HIV Infections; Histoplasmosis; Acquired Immunodeficiency Syndrome; Recurrence | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To evaluate the use of fluconazole as (1) induction therapy in histoplasmosis, (2) maintenance therapy to prevent relapse of histoplasmosis.

Histoplasmosis is a serious opportunistic infection in patients with AIDS. Fluconazole is a triazole antifungal agent that has been used successfully in the treatment of experimental histoplasmosis in animals, but has not been completely evaluated in patients for this use. It has been approved by the Food and Drug Administration for certain other fungal infections. Nevertheless, physicians are prescribing it to their patients with histoplasmosis. This is a pilot study to examine the role of fluconazole for treating histoplasmosis in AIDS patients.

DETAILED DESCRIPTION:
Histoplasmosis is a serious opportunistic infection in patients with AIDS. Fluconazole is a triazole antifungal agent that has been used successfully in the treatment of experimental histoplasmosis in animals, but has not been completely evaluated in patients for this use. It has been approved by the Food and Drug Administration for certain other fungal infections. Nevertheless, physicians are prescribing it to their patients with histoplasmosis. This is a pilot study to examine the role of fluconazole for treating histoplasmosis in AIDS patients.

At least 40 patients with AIDS and an initial episode of disseminated histoplasmosis are selected for the study. Patients receive fluconazole for a total of 12 weeks. Patients who are unable to take the drug orally may receive it intravenously until oral administration is possible. Patients are evaluated at weeks 0, 1, 2, 4, 8, and 12. Patients who are doing well without evidence of clinical failure or dose-limiting toxicity are permitted to continue maintenance therapy to prevent relapse at a reduced dose for an additional 12 months; those who relapse on the reduced dose are permitted to receive re-induction with a higher dose.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Corticosteroids for up to 21 days at doses no greater than 20 mg/day prednisone (higher doses may be given for shorter durations, if clinically indicated).
* Zidovudine, oral contraceptives, methadone, narcotics, acyclovir, acetaminophen, sulfonamides, trimethoprim/sulfamethoxazole, pentamidine for Pneumocystis carinii pneumonia (PCP) or PCP prophylaxis, topical antifungals, pyrimethamine, ganciclovir.
* Didanosine (ddI), dideoxycytidine (ddC), foscarnet, or other investigational drugs considered to be essential for patient management.

Concurrent Treatment:

Allowed:

* Transfusion.

Patients must have the following:

* HIV infection.
* Histoplasmosis.
* Appropriate consent must be obtained from a parent or legal guardian for patients less than 18 years of age.

Allowed:

* Hematologic and/or renal laboratory abnormalities.
* Concurrent malignancies.
* Concurrent infection with Mycobacteria.
* Patients with severe manifestations of histoplasmosis who are thought to be at risk of dying within one week should receive up to 250 mg amphotericin B for up to seven days prior to enrollment and then be re-evaluated. Patients who are still severely ill and do not meet eligibility criteria may not enter the study.

Specific criteria defining life-threatening histoplasmosis include:

* Systolic blood pressure < 90 mm Hg without other cause; arterial pO2 < 60 torr without other cause; and SGOT > 10 x upper limit of normal or bilirubin > 3 x upper limit of normal. Any other cases not meeting this definition must be reviewed with the protocol chair.

Prior Medication:

Allowed:

* Amphotericin B (up to 250 mg) over 7 days in patients with severe histoplasmosis.

Risk Behavior:

Allowed:

* Patients with a history of high-risk behavior for HIV infection (bisexual or homosexual men, intravenous drug abusers, recipients of blood or blood products prior to May 1985, or sexual partners of any of the foregoing).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Allergy to, or intolerance of, imidazoles or azoles.
* Active hepatitis (viral, drug induced, or other).
* Fungal infections for which the study drug is not indicated (e.g., aspergillosis, mucormycosis).
* CNS/CSF culture positive for pathogens other than H. capsulatum. If C. neoformans is subsequently identified and the patient is improving, the patient may be allowed to remain on study with the permission of the protocol chair.

Concurrent Medication:

Excluded:

* Corticosteroid use for > 21 days at > 20 mg/day of prednisone.
* Systemic antifungals.

Prior Medication:

Excluded:

* Amphotericin B at > 2.5 mg/kg for the current episode of histoplasmosis within 7 days prior to enrollment.
* Suppressive treatment for histoplasmosis or other fungal infections with > 200 mg/day of ketoconazole, fluconazole, or itraconazole, or more than 50 mg amphotericin B twice weekly.

Risk Behavior:

Excluded:

* Patients who the investigator feels would be undependable with regard to adherence to the protocol.

Patients may not have the following prior conditions:

* History of allergy to, or intolerance of, imidazoles or azoles.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Study Completion 1994-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wheat LJ, Study Chair
Locations (23):
- United States (23):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Worcester Memorial Hosp / Med Ctr of Cntrl MA-Memorial, Worcester, Massachusetts
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Infectious Diseases Association / Research Med Ctr, Kansas City, Missouri
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Beth Israel Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas

REFERENCES:
- [Background] Wheat J, Vanden Bossche H, Marichal P. Mechanism for resistance of Histoplasma capsulatum to fluconazole. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:157
- [Background] Wheat J, MaWhinney S, Hafner R, McKinsey D, Chen D, Korzun A, Shakan KJ, Johnson P, Hamill R, Bamberger D, Pappas P, Stansell J, Koletar S, Squires K, Larsen RA, Cheung T, Hyslop N, Lai KK, Schneider D, Kauffman C, Saag M, Dismukes W, Powderly W. Treatment of histoplasmosis with fluconazole in patients with acquired immunodeficiency syndrome. National Institute of Allergy and Infectious Diseases Acquired Immunodeficiency Syndrome Clinical Trials Group and Mycoses Study Group. Am J Med. 1997 Sep;103(3):223-32. doi: 10.1016/s0002-9343(97)00151-4. PMID 9316555